CLINICAL TRIAL: NCT04927377
Title: Accessible and Inclusive Diabetes Telecoaching Self-Management Program: Protocol for a Feasibility Study
Brief Title: Accessible and Inclusive Diabetes Telecoaching Self-Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-300007168
Record Dates: First submitted 2021-06-04; First posted 2021-06-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Diabete Type 2; Disability Physical
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The principal investigator and biostatistician will be masked to the randomization of the participants into the two treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI4DM Intervention Group (Experimental)
  Interventions: Behavioral: AI4DM
- Attention-control Group (Active Comparator)
  Interventions: Behavioral: Attention-control

INTERVENTIONS:
Behavioral: AI4DM — Those in the AI4DM intervention arm will receive weekly and bi-weekly calls for six months, access to home and online technology, diabetes-related multimedia educational content, a technology package including a voice-assistive device, wireless glucometer, and wrist-worn activity monitor
  Arms: AI4DM Intervention Group
Behavioral: Attention-control — Those in the Attention-control Group will receive telecoaching calls at the same frequency of the Intervention Group. Coaching calls will focus on general wellbeing, rather than diabetes-related topics. The Attention-control Group will serve as an untreated comparison group for the Intervention Group.
  Arms: Attention-control Group

SUMMARY:
The purpose of this study is to develop and pilot test an accessible and inclusive Artificial Intelligence (AI)-assisted, individualized, family-focused lifestyle modification intervention (AI4DM) for glycemic control in people with disabilities.

DETAILED DESCRIPTION:
The AI4DM study will use a two-arm randomized control trial design. Eligible and consented participants will be assigned to one of two groups: 1) AI4DM intervention group with telecoaching support, and 2) attention-control group. The active intervention period will include six months of weekly and bi-weekly telecoaching calls followed by six months of follow-up and technology access, but no telecoaching calls.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus,
* Living with a permanent physical disability such as spinal cord injury (SCI), spina bifida, multiple sclerosis, stroke, etc.
* Ability to converse and read in English

Exclusion Criteria:

* Current enrollment in any diabetes-related intervention
* Severe untreated depression in the past six months
* Major cardiac event in the past twelve months
* Uncontrolled blood pressure
* Resting tachycardia
* Renal failure
* Severe peripheral neuropathy
* Unavailability of a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Glycemic Management | 48 weeks
  Measured using HbA1c

SECONDARY OUTCOMES:
Psychological distress | 48 weeks
  Measured using Diabetes Distress Scale (DDS); Minimum score = 1, maximum score = 6; Higher score represents worse outcome
Diabetes Quality of life | 48 weeks
  Measured using the DQoL (Diabetes Quality of Life Measure) Questionnaire; Minimum score =1; maximum score = 5; Higher score represents worse outcome
Self-efficacy | 48 weeks
  Measured using Diabetes Empowerment Scale; Minimum score = 1; maximum score = 5; Higher score represents better outcome
Family Support | 48 weeks
  Measured using the Diabetes Social Support Questionnaire - Family Version (DSSQ-Family); Minimum score = -5 maximum score = 15; Higher score represents better outcome
Physical Activity | 48 weeks
  Measured using Godin leisure-time exercise questionnaire; Minimum score = 0; Maximum score = unknown; Higher score represents better outcome
Dietary intake | 48 weeks
  Measured using The UK Diabetes and Diet Questionnaire
Medication Adherence | 48 weeks
  Measured using the Medication Adherence Rating Scale
Health Information Technology | 48 weeks
  Measured using The eHealth Literacy Scale
Telehealth Dashboard Usability | 48 weeks
  Measured using the System Usability Scale; Maximum item score (Strongly agree) = 5, minimum item score (Strongly disagree) = 1; Higher scores represent better outcomes
Health Technology Usability | 48 weeks
  Measured using the Health Information Usability Evaluation Scale (Health-ITUES)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be submitted to ICPSR.
Supporting Information: Analytic Code

REFERENCES:
- [Background] Wolff K, Chambers L, Bumol S, White RO, Gregory BP, Davis D, Rothman RL. The PRIDE (Partnership to Improve Diabetes Education) Toolkit: Development and Evaluation of Novel Literacy and Culturally Sensitive Diabetes Education Materials. Diabetes Educ. 2016 Feb;42(1):23-33. doi: 10.1177/0145721715620019. Epub 2015 Dec 7. PMID 26647414
- [Background] Ali MK, Echouffo-Tcheugui J, Williamson DF. How effective were lifestyle interventions in real-world settings that were modeled on the Diabetes Prevention Program? Health Aff (Millwood). 2012 Jan;31(1):67-75. doi: 10.1377/hlthaff.2011.1009. PMID 22232096
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Derived] Zengul A, Evans E, Hall A, Qu H, Willig A, Cherrington A, Thirumalai M. Telehealth Behavioral Intervention for Diabetes Management in Adults With Physical Disabilities: Intervention Fidelity Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Sep 10;10(9):e31695. doi: 10.2196/31695. PMID 34505835
- [Derived] Evans E, Zengul A, Hall A, Qu H, Willig A, Cherrington A, Thirumalai M. Disability-Inclusive Diabetes Self-management Telehealth Program: Protocol for a Pilot and Feasibility Study. JMIR Res Protoc. 2021 Sep 10;10(9):e31689. doi: 10.2196/31689. PMID 34505831